CLINICAL TRIAL: NCT02074644
Title: Randomized, Evaluator-blind, Controlled Trial to Evaluate the Efficacy and Safety of Prostatic Arterial Embolization Versus a Sham Procedure for Benign Prostatic Hyperplasia With Severe LUTS Not Adequately Controlled With Alpha-blockers
Brief Title: Clinical Trial of Prostatic Arterial Embolization Versus a Sham Procedure to Treat Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: João Martins Pisco (Other)
Responsible Party: Sponsor-Investigator, João Martins Pisco, Professor, Hospital St. Louis, Lisbon, Portugal
Organization: Hospital St. Louis, Lisbon, Portugal (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAE-01-2013
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Prostatic Hyperplasia, Benign; Prostatic Hypertrophy, Benign; Genital Diseases, Male; Lower Urinary Tract Symptoms; Prostatic Diseases
Keywords: Prostatism; Randomized Controlled Trial; Embolization, Therapeutic; Hyperplasia; Prostatic Diseases; Genital Diseases, Male
MeSH Terms: conditions — Prostatic Hyperplasia; Genital Diseases, Male; Lower Urinary Tract Symptoms; Prostatic Diseases; Prostatism; Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostatic Arterial Embolization (Experimental): Selective catheterization of the prostatic arteries followed by slow injection of Bead Block 300-500 or PVA 100+200 micra particles under fluoroscopic control.
  Interventions: Procedure: Prostatic Arterial Embolization
- Sham procedure (Sham Comparator): Selective catheterization of the prostatic arteries followed by removal of the catheter with no particles injected.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Prostatic Arterial Embolization — The prostatic arteries are selectively catheterized with a Progreat 2.7 microcatheter and an angiography is performed to confirm that the catheter is in the prostatic artery. Bead Block 300-500 or PVA 100+200 micra particles are slowly injected under fluoroscopic control until the end point is reached. Embolization is considered finished when there is "near stasis" in the prostatic vessels with interruption of the arterial flow and prostatic gland opacification checked in both oblique and AP views. Upon finishing the embolization of the left prostatic arteries, the right prostatic arteries are embolized in the same way.
  Arms: Prostatic Arterial Embolization
Procedure: Sham procedure — The prostatic arteries are selectively catheterized with a Progreat 2.7 microcatheter and an angiography is performed to confirm that the catheter is in the prostatic artery. The catheter is removed and no particles are injected.
  Arms: Sham procedure

SUMMARY:
The purpose of this study is to determine whether prostatic arterial embolization (PAE) compared is an effective and safe treatment for benign prostatic hyperplasia in patients with severe lower urinary tract symptoms not adequately controlled by medical therapy with alpha-blockers, as assessed by the the International Prostate Symptom Score (IPSS) after 6 months. Patients will be randomized on a 1:1 ratio to PAE or to a sham procedure and evaluated at 1, 3 and 6 months. Patients randomized to the sham procedure will be offered the possibility of performing PAE after 6 months. All patients may participate on an optional 6-months extension study.

DETAILED DESCRIPTION:
This is a randomized, parallel-group, evaluator-blind, superiority, controlled clinical trial of PAE versus a sham procedure in patients with BPH with severe LUTS not adequately controlled by medical therapy with alpha-blockers.

This study has a screening visit at day -14, a baseline visit at day -2, a randomization and intervention visit at day 0, follow up visits at months 1, 3 and 6.

Patients initially randomized to the sham procedure and who completed the 6 month follow-up period will be offered the possibility of performing PAE at no cost. All patients will be invited to participate in a 6 months post-trial extension study.

Patients over 45 years-old with a diagnosis of BPH associated with severe LUTS defined by an IPSS>=20 after a minimum of 6 months treatment with alpha-blockers and with a prostate volume ≥ 40 mL will start a two weeks screening period. Eligible patients will be started either tamsulosin 0.4 mg q.d., alfuzosin 10 mg q.d. or silodosin 8 mg q.d., which will be maintained throughout the study period, and have the intervention scheduled for the following 2 days (study day 0), when they will be randomized to PAE or to a sham procedure if the procedure is technically feasible

Those patients in whom angiography has shown that PAE is technically feasible will be randomized to one of the study arms on a 1:1 ratio. Patients in both groups will be submitted to exactly the same procedure, except that patients randomized to the control group will not be injected with polyvinyl alcohol particles. Patients will be discharged as soon as their clinical condition is stabilized

Patients will be assessed at 1, 3 and 6 months with IPSS, QoL, IIEF, BPH-II and will perform prostatic ultrasonography, uroflowmetry and PSA at month 1 and 6. At 1 month a pelvic NMR will be performed to evaluate prostate volume and the degree of ischemia.

Patients completing the 6 month follow-up period will be invited to enter a 6 months extension study. In this extension study, patients will be evaluated at month 12 for all efficacy variables. Patients initially randomized to the sham procedure who wanted to perform PAE after the conclusion of the trial will be evaluated only at months 1, 3 and 6 after PAE.

ELIGIBILITY:
Inclusion Criteria:

* Male patients ≥ 45 years-old
* Diagnosis of BPH based on clinical history, digital rectal examination, urine sediment, transrectal prostate ultrasound and PSA
* Use of a marketed alpha-blocker for LUTS/BPH in the previous 6 months
* Severe lower urinary tract symptoms at screening and baseline defined by all the following: IPSS (7 items) ≥ 20, QoL ≥ 3, Qmax < 12 mL/s and prostate volume ≥ 40 mL
* CTA shows that prostatic arteries are feasible for PAE
* Sexual dysfunction or accepting the risk of developing sexual dysfunction after treatment
* Written informed consent

Exclusion Criteria:

* Previous surgical or invasive prostate treatments such as TURP, TUMT, TUNA, laser or any other minimally invasive treatment
* Acute or chronic prostatitis or suspected prostatitis including chronic pain, intermittent pain or abnormal sensation in the penis, testis, anal or pelvic area in the past 12 months
* History of prostate or bladder cancer or pelvic irradiation
* Active or recurrent urinary tract infections (more than 1 episode in the last 12 months)
* History of neurogenic bladder or LUTS secondary to neurological disease
* Advanced atherosclerosis and tortuosity of iliac and prostatic arteries
* Secondary renal insufficiency (due to prostatic obstruction)
* Large bladder diverticula or stones
* Detrusor failure
* Previous history of acute urinary retention
* Current severe, significant or uncontrolled disease (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal, uncontrolled hypertension (systolic ≥ 160 mmHg and/or diastolic ≥95 mmHg), congestive heart failure [New York Heart Association status of class III or IV], myocardial infarction within 26 weeks prior to randomization), which in the judgment of the clinical investigator renders the subject unsuitable for the trial and puts the subject at increased risk
* Any bleeding disorder such as hemophilia, clotting factor deficiency, anti-coagulation or bleeding diathesis
* Hypersensitivity or contraindication to tamsulosin use
* Administration of 5-ARIs, finasteride and dutasteride in the previous 2 weeks and 4 months, respectively. These patients may be included if they stop those medications and replace them for tansulosin, alfuzosin or silodosin for at least 2 weeks and 4 months, respectively.
* Any mental condition or disorder that would interfere with the subject's ability to provide informed consent
* Participation in a study of any investigational drug or device in the previous 3 months

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the International Prostate Symptom Score | 6 months
  The difference between the baseline value and the value observed at the last valid observation of a validated questionnaire that measures the disconfort caused by lowere urinary tract symptoms

SECONDARY OUTCOMES:
Disease specific quality of life question of the International Prostate Symptom Score | 6 months
  The score of a question on the IPSS questionnare that measures quality of life in subjects with lower urinary tract symptoms at the last valid observation in each subject

OTHER OUTCOMES:
Change from baseline in the Benign Prostatic Hyperplasia Impact Index (BPH-II) | 6 months
  The difference between the baseline value and the value observed at the last valid observation on a validated questionnaire that measures the disconfort caused by lowere urinary tract symptoms
Change from baseline in the International Index of Erectile Function (IIEF) | 6 months
  The difference between the baseline value and the value observed at the last valid observation on a validated questionnaire that measures the severity of erectile disfunction
Change from baseline in the peak urinary flow rate (Qmax) | 6 months
  The difference between the baseline value and the value observed at the last valid observation of the maximum flow rate of the urinary stream by uroflowmetry
Change from baseline in the post-void residual volume | 6 months
  TThe difference between the baseline value and the value observed at the last valid observation of he volume of urine in the bladder after a complete voiding assessed by uroflowmetry
Change from baseline in prostate volume | 6 months
  The difference between the baseline value and the value observed at the last valid observation of prostate volume measured by transrectal ultrasonography
Change from baseline in the Prostate Specific Antigen (PSA) | 6 months
  The difference between the baseline value and the value observed at the last valid observation of PSA.

CONTACTS AND LOCATIONS:
Overall Officials: João M Pisco, M.D,. Ph.D., Study Director — Hospital de Saint Louis
Locations (1):
- Hospital de Saint Louis, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary of all the study data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From January 2020
Access Criteria: Deidentified participant data and data dictionary will be made available upon request to oliveira.amg@gmail.com with the submission of a study protocol and subsequent approval by the Research Ethics Committee of the institution where the trial was conducted.

REFERENCES:
- [Result] Pisco JM, Bilhim T, Costa NV, Torres D, Pisco J, Pinheiro LC, Oliveira AG. Randomised Clinical Trial of Prostatic Artery Embolisation Versus a Sham Procedure for Benign Prostatic Hyperplasia. Eur Urol. 2020 Mar;77(3):354-362. doi: 10.1016/j.eururo.2019.11.010. Epub 2019 Dec 10. PMID 31831295